CLINICAL TRIAL: NCT07044869
Title: Effects of Facilitated Positional Release Technique( FPRT) Vs Manual Myofascial Release Technique in Female Patients With Piriformis Syndrome.
Brief Title: Effects of Facilitated Positional Release Technique ( FPRT) Vs Manual Myofascial Release Technique in Female Patients With Piriformis Syndrome.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/81
Record Dates: First submitted 2025-06-01; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Piriformis Syndrome
MeSH Terms: conditions — Piriformis Muscle Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Positional Release group (Active Comparator): On group A we will perform FACILITATED POSITIONAL RELEASE TECHNIQUE:
  we perform this technique on tight PIRIFORMIS muscle.
  Interventions: Procedure: FACILITATED POSITIONAL RELEASE TECHNIQUE
- Group B Myofascial release group (Experimental): On group B we perform MANUAL MYOFASCIAL RELEASE TECHNIQUE on tight PIRIFORMIS muscle same as group A
  Interventions: Procedure: MANUAL MYOFASCIAL RELEASE TECHNIQUE

INTERVENTIONS:
Procedure: FACILITATED POSITIONAL RELEASE TECHNIQUE — Participants in experimental group A receive FPRT as a main intervention along with piriformis stretches. 30 minutes' session starts with application of 10 minutes hot pack, followed by FPRT and stretches respectively. For FPRT, the patient position was prone with the hip flexion approximately (60°-90°) and abduction. The therapist was seated on the side that was affected, and the treated leg was hanging off the table with the knee bent resting on the therapist thigh. The painful tender area was felt in the piriformis muscle's belly around midway between the greater trochanter and the inferior lateral angle of sacrum. At the point when tender area was palpated, therapist applied ischemic pressure over the area with finger pads. Pressure hold for 1 minute and two repetitions were performed (2 minutes' pressure for whole was given). After that piriformis stretches were performed with 5reps*5 sec hold*1set.
  Arms: Group A Positional Release group
Procedure: MANUAL MYOFASCIAL RELEASE TECHNIQUE — Experimental Group B participants received MFRT as a main intervention along with application of hot pack and piriformis stretches. They also received 30 min session started with application of hot pack for 10 minutes followed by MFRT and piriformis stretches. For application of MFRT patient was in prone lying position. The therapist was standing at the affected/unaffected side of the patient. Myofascial release was provided, using the therapist's palm, finger pads or elbow directly on the piriformis muscle, pressure was provided on the tender area directly and held for a while (60 seconds approx.) and 3 repetitions were performed. Back and forth little kneading motions were applied in accordance with the muscle fiber's direction. After MFRT piriformis stretches were performed with frequency of 5 repetitions *5 second hold* 1 set.
  Arms: Group B Myofascial release group

SUMMARY:
This study is a randomized control trial, and the purpose of this study is to determine the "Effects of Facilitated Positional Release Technique ( FPRT) Vs Manual Myofascial Release Technique in Female Patients with Piriformis Syndrome.

DETAILED DESCRIPTION:
The purpose of this study is to determine the "Effects of Facilitated positional release technique vs manual myofascial release technique in female patietns with piriformis syndrome.

we make 2 groups control and treatment group . we give FPRT technique to treatment group and manual release technique to control group in patients with piriformis syndrome.

first we take base line readings of HIP ROMS( abduction, adduction, internal rotation, external rotation),NPRS and LEFS(lower extremity functional scale)..

after 2 weeks of treatment again we take same readings and compare both readings.

ELIGIBILITY:
Inclusion Criteria:

* • 25-50 years Only females Diagnosed piriformis syndrome Pain from 2 months

Exclusion Criteria:

* Lumbar Radiculopathy Fracture trauma to lumbar spine surgery/ total hip replacement hip OA

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 25 to 50 years females suffering from piriformis syndrome
Enrollment: 38 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Piriformis Pain | Before and after every 2 sessions for a total of 2 weeks
  The NPRS which has eleven points ranging from zero (0) to ten (10) is used to quantify the degree of pain before and after. A score of 0 denotes "no pain", while score of 10 denotes: maximally felt pain".
Lower Extremity Functional Scale | Before and after every 2 sessions for a total of 2 weeks
  Lower extremity functional scale consisting of 20 questions about lower extremity function is used. The highest possible count is 80 points, indicating greatest function. The least possible count is 0 points, indicating poor function.
Range of Motion | Before and after every 2 sessions for a total of 2 weeks.
  The ranges of hip abduction, hip adduction, hip internal and external rotations are measured using goniometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan